CLINICAL TRIAL: NCT02259062
Title: Measuring the Effects of Listening for Leisure on Outcome After Stroke (MELLO)
Brief Title: Listening for Leisure After Stroke
Acronym: MELLO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GN13CP462
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Music listening (Active Comparator)
  Interventions: Other: Music listening alone
- Music listening with brief mindfulness (Experimental)
  Interventions: Other: Music with brief mindfulness intervention
- Audio book intervention (Placebo Comparator)
  Interventions: Other: Audiobook listening

INTERVENTIONS:
Other: Music with brief mindfulness intervention — Music listening with mindfulness therapy
  Arms: Music listening with brief mindfulness
Other: Music listening alone
  Arms: Music listening
Other: Audiobook listening
  Arms: Audio book intervention

SUMMARY:
Stroke is the biggest cause of disability in older adults. Early poststroke rehabilitation focuses primarily on physical disability and activities of daily living. By contrast, relatively little research attention has been paid to the potential for cognitive rehabilitation and mood enhancing interventions in the early stages after stroke. Low mood and cognitive difficulties with attention and memory are common post stroke leading to poorer recovery, emotional wellbeing and quality of life yet accessible and effective therapies are lacking.

Engagement in leisure activities may enhance recovery after stroke but participation in leisure activities is reduced following stroke. Music listening is a low cost and accessible leisure activity that has been suggested to improve mood and cognition poststroke. The investigators speculate that music listening may enhance control of attention in a similar way to mindfulness interventions, that have been demonstrated to be beneficial in the treatment of mood disorders. The investigators propose that adding a brief mindfulness intervention to music listening might enhance the effect on control of attention, with positive effects on cognition and mood poststroke but the feasibility and acceptability of this intervention needs to be evaluated before attempting a further trial assessing the effectiveness of this intervention. The investigators aim to recruit 100 patients within two weeks poststroke.

Participants will be randomly assigned to receive an 8 week music listening alone, music listening with brief mindfulness or audiobook listening intervention alongside treatment as usual. Neuropsychological assessment of cognition and mood will be performed at baseline, 3 months, and 6 months poststroke In addition, participants will be interviewed about their experience of engaging in the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ischaemic stroke (confirmed clinically and/or radiologically and subclassified according to the Oxford Clinical Stroke Classification)
* ≤14 days poststroke at time of recruitment (expression of interest to participate either verbally or in writing)
* Native English speaking

Exclusion Criteria:

* Comorbid progressive neurological or neurodegenerative condition
* Major psychiatric disorder (Prestroke history of mood disorder or stable antidepressant medication will not lead to exclusion)
* History of major substance abuse problems
* Unable to give informed consent
* Unable to cooperate with the study protocol (e.g. due to severe aphasia, uncorrected impairment of hearing or vision, or illiteracy)
* Clinically unstable (e.g. due to major intercurrent illness).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate at 6 month follow up from baseline | 6 months
Treatment adherence at 6 month follow up from baseline | 6 months
sample retention at 6 month follow up from baseline | 6 months

SECONDARY OUTCOMES:
Change in overall cognition score at 6 months from baseline | 6 months
Change in attention, memory and executive function scores at 6 months from baseline | 6 months
Change in Hospital Anxiety and Depression Scale (HADS) scores at 6 months from baseline | 6 months
Changes in Five Facet Mindfulness Questionnaire short form (FFMQ-sf) | 6 months
Changes in Mayo Portland Adaptability Inventory 4 (MPAI-4) scores | 6 months
Changes in Brain Injury Rehabilitation Trust Regulation of Emotions Adaptability | 6 months
Changes in Metacognitions Questionnaire short form (MCQ-30) | 6 months
Likert ratings of participants' and therapist's experiences of treatment delivery. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Evans, BSc,Dip.Clin.Psychol. PhD, Principal Investigator — University of Glasgow
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom